CLINICAL TRIAL: NCT02282800
Title: Immunolocalization of 1,25,Dihydroxyvitamin D3 in Aggressive Periodontitis Patients
Acronym: IVDAP
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.Dasari Rajashre, Immunolocalization of 1,25,Dihydroxyvitamin D3 in Aggressive Periodontitis Patients, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: PanineeyaMVIDS
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Receptors, Calcitriol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group: Case group include patients with generalized AgP were the tissue samples taken to analyse the number of vitamin D receptor present.
  Interventions: Genetic: Vitamin D receptor
- Control group: Ethnically matched, systemically and periodontally healthy individuals were included in control group were also gingival tissue taken for analysis of number of receptors present in nucleus and cytoplasm
  Interventions: Genetic: Vitamin D receptor

INTERVENTIONS:
Genetic: Vitamin D receptor — 50-100mg gingival tissue samples were collected from both test and control group for immunohistochemical staining to assess the number of vitamin D receptors in nucleus as well cytoplasm and also for RNA isolation to check the presence of VDR gene.
  Other Names: 1,25,dihydroxyvitamin D3 receptor

SUMMARY:
The study was to intended to visualize the nuclear localization of vitamin D receptor in oral tissues of aggressive periodontitis patients to better understand the potential for receptor in disease activity or progression.

DETAILED DESCRIPTION:
Aggressive periodontitis (AgP) is an infectious disease of the periodontium which affects young adults, causing damage to the supporting apparatus of the teeth, leading to rapid bone resorption and tooth loss. Its clinical features have been shown to result from several genetic and environmental factors.

This has increased the interest to research those genetic host factors as they may provide useful risk markers, reveal important information regarding the pathogenesis and also identification of effective preventive agents that might help decrease the disease burden.

1,25-dihydroxyvitamin D3,apart from these traditional calcium-related actions, this active form is being increasingly recognized for its potent anti-proliferative, anti-differentiative and immunomodulatory activities.

The calcitriol activity is largely mediated by the vitamin D receptor (VDR) whose expression has been described in some tissues. VDR is localized in both the cytosol and nucleus and accumulates in the nucleus in response to 1,25,dihydroxyvitamin D3 binding.

Expression and nuclear activation of the VDR are necessary for the effects of vitamin D. Thus, alterations in the vitamin D pathway lead to disturbances in mineral metabolism. It may be hypothesized that the rapid bone loss which occurs in aggressive periodontitis patients may be due to decreased or absence of expression of Vitamin D receptor in the nucleus.

ELIGIBILITY:
Inclusion Criteria:

1. Generalized Aggressive periodontitis patients were onset of periodontal disease at <35yrs of age and atleast eight teeth with probing depth >6mm and radiographic evidence of alveolar bone loss, three of which were not first molar or incisor under test group.
2. Control group includes systemically and periodontally healthy individuals who is of same age as that of test group.

   -

Exclusion Criteria

1. Subjects taking drugs for vitamin D or calcium
2. Subjects received periodontal therapy within previous year
3. Pregnant subjects
4. Smokers
5. Patients with systemic diseases -

Ages: 24 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population was divided in to two groups i.e test and control group
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Less nuclear receptors in aggressive periodontitis | 24hrs
  Immunohistochemical staining has been done for test group and control group tissue samples where less nuclear vitamin D receptors are found in aggressive periodontitis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rajashree Dasari, MDS, Principal Investigator — Panineeya Mahavidyalaya